CLINICAL TRIAL: NCT01884142
Title: Effects of Exercise Training on Mechanoreflex and Metaboreflex Control of Muscle Sympathetic Nerve Activity in Heart Failure Patients
Brief Title: Effects of Exercise Training on Mechanoreflex and Metaboreflex Control in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Lígia M. Antunes-Correa, PhD student, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ergoreflex
Record Dates: First submitted 2013-03-27; First posted 2013-06-21 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heart Failure Untrained Group (No Intervention): Control Group
- Heart Failure Exercise-trained Group (Experimental): Aerobic Exercise Training
  Interventions: Other: Aerobic Exercise Training

INTERVENTIONS:
Other: Aerobic Exercise Training
  Arms: Heart Failure Exercise-trained Group

SUMMARY:
The investigators hypothesize that exercise training would improve the mechanoreflex and metaboreflex control in heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with systolic heart failure;
* New York Heart Association (NYHA) class II-III;
* Left ventricular ejection fraction less than 40%;
* Peak Oxygen Consumption less than 20 ml/Kg/min;
* Stable Clinical Status.

Exclusion Criteria:

* Chronic Obstructive Pulmonary Disease;
* Neuromuscular Diseases;
* Orthopedic Diseases;
* Neurologic Diseases;
* Neoplastic Diseases;
* Recent myocardial infarction or cardiac surgery (less than 6 months);
* Unstable angina pectoris;
* Atrial Fibrillation;
* Pacemakers users;
* Changing medication or hospital admission.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Autonomic Control | 4 months
  Mechanoreceptors were activated by passive exercise and metaboreceptors by post-exercise circulatory arrest
Muscular Evaluation | 4 months
  Muscular evaluation will be done by muscle gene expression

SECONDARY OUTCOMES:
Functional Capacity | 4 months
  Functional Capacity will be determined by cardiopulmonary exercise testing
Muscle Blood Flow | 4 months
  Forearm blood flow will be assessed by venous occlusion plethysmography
Blood Pressure | 4 months
  Blood pressure will be monitored non-invasively

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Negrão, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Heart Institute (InCor), University of Sao Paulo Medical School, São Paulo, Brazil

REFERENCES:
- [Background] Unable to connect to PubMed to validate , last attempt on June 19, 2013 at 12:03 PM EDT